CLINICAL TRIAL: NCT04358042
Title: PSYCHIatric Disorders and Covid-19 (PSYCHIC) : Observatory of the Psychiatric, Somatic and Pharmacological Impacts of the COVID-19 Pandemic on Patients Hospitalized for Psychiatric Disorders and Suspected to be Infected by COVID-19
Brief Title: PSYCHIATRIC Disorders and Covid-19
Acronym: PSYCHIC
Status: Terminated | Type: Observational
Why Stopped: Impossibility of recruitment because Covid service not renewed.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0165
Record Dates: First submitted 2020-04-08; First posted 2020-04-22 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Psychiatric Disorder; Covid19
Keywords: Psychiatry; COVID-19; psychological impact; acute stress, pharmacological impact; pharmacological impact
MeSH Terms: conditions — Mental Disorders; COVID-19 | interventions — Brief Psychiatric Rating Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Brief Psychiatric Rating Scale — The Abbreviated Psychiatric Rating Scale is a clinical scale for measuring symptomatic change in psychiatric inpatients for various conditions. It includes an accurate and complete description of the major characteristic symptoms. It is based both on patient responses and on observations made during the interview by the clinician. The usual reference period is the last two weeks.
Other: Depression, Anxiety and Stress Scale — evaluation of 3 dimensions of psychological distress: depression, anxiety and stress. The scale consists of 21 items and the patient is instructed to choose for each item the one that best corresponds to his or her experience over the past week, on a scale of 0 ("does not apply to me at all") to 3 ("applies entirely to me, or the vast majority of the time"). A score is calculated for each dimension according to a predefined rating.
Other: Impact of Event Scale-Revised — is a 22-item self-questionnaire that measures perceived stress in reference to a traumatic event during the previous 7 days. Each item is rated on a scale ranging from 0 (not at all) to 4 (extremely) and 3 sub-scores of post-traumatic symptoms are calculated: Revivification, Avoidance, Psychophysiological Activation, as well as a total score of severity of the state of stress. Acute Stress Disorder (ASD) and Post-Traumatic Stress Disorder (PTSD) share the same symptoms, the former lasting between 3 days and one month, while the latter is diagnosed when symptoms persist beyond one month. Since the exposure to the stressful event will have occurred less than a month ago, this questionnaire here will help identify a state of acute stress. A total R-ESI score equal to or greater than 33 suggests a significant level of symptoms
Other: Connor-Davidson Resilience Scale 10 items (CD-RISC 10) — Self-questionnaire composed of 10 items, evaluating the resilience capacities of patients. Resilience may act as a moderator against the symptoms of PTSD. This instrument uses a 5-point Likert-type response scale ranging from 0 "Not true at all" to 4 "True most of the time".

SUMMARY:
Given the possible risks and complications of a comorbidity between psychiatric disorder and coronavirus disease 2019 (COVID-19), it seems particularly important to specify the impact of the COVID-19 pandemic in patients with psychiatric disorders and suspected of infection, hospitalized in a specific unit, at the psychiatric, somatic and pharmacological level.

DETAILED DESCRIPTION:
COVID-19's possible impact on psychiatric disorders has been little studied. However, patients with psychiatric disorders may be at higher risk of COVID-19 contamination, may experience delayed treatment when infected, may have a poor prognosis in terms of complications and success of treatment for COVID-19 but also for the underlying psychiatric disorder which could be exacerbated, and finally their psychotropic pharmacological treatment could be impacted by the inflammatory state linked to COVID-19.

The present study is an observatory of patients with psychiatric disorders and suspected to be infected by the COVID-19, hospitalized in a specific unit dedicated to the treatment of this comorbidity in the University Hospital of Nantes (France). The primary objective is to investigate the impact of the COVID-19 pandemic on the level of acute traumatic stress response. Secondary objectives include: (i) a description of the sample included; (ii) an assessment of the clinical evolution of these patients 4-6 weeks after admission; (iii) to investigate the links between the levels of stress, peritraumatic distress, and traumatic stress (whether it is acute or has evolved into a post-traumatic stress disorder (PTSD)); (iv) to investigate the links between resilience and coping on the one hand, and stress, peritraumatic distress and traumatic stress (acute or PTSD) on the other hand; and (v) to measure the impact of COVID infection and of the reduction on the residual plasma concentrations of psychotropic medications (especially antipsychotics and lithium).

ELIGIBILITY:
Inclusion Criteria:

* All patients hospitalized in the PROTECTION COVID-19 PSY unit from the Nantes University Hospital may be included, without maximum age limit.

Minors, pregnant or nursing women, and patients under guardianship and tutorship may be included, taking into account the study population and the low risks and constraints of the study (observatory)

Exclusion Criteria:

* minors under 15 years;
* safeguard of justice;
* inability to consent (non-opposition);
* not mastering the reading and writing of the French language well enough.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with psychiatric disorders and suspected to be infected by the COVID-19, hospitalized in a specific unit dedicated to the treatment of this comorbidity in the University Hospital of Nantes (CHU Nantes).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
impact of the COVID-19 pandemic on psychiatric symptomatology | through study completion, an average of 2 year
  total severity score from the Impact of Event Scale-Revised (IES-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital - IFAC, Nantes, Loire-Atlantique, France